CLINICAL TRIAL: NCT06706973
Title: Profiling and Targeting Epigenetic Marks to Improve Diagnosis and Therapeutic Approaches in Head and Neck Cancer
Acronym: AIRC-Chiocca
Status: Recruiting | Type: Observational
Sponsor: European Institute of Oncology (Other)
Collaborators: AIRC (Italian Association for Cancer Research) (Unknown)
Responsible Party: Sponsor
Other Study IDs: IEO 1972
Record Dates: First submitted 2024-11-22; First posted 2024-11-27 (Actual); Last update posted 2024-11-27 (Actual); Status verified 2024-10

CONDITIONS: Head and Neck Cancer
Keywords: PROFILING AND TARGETING EPIGENETIC MARKS; HEAD AND NECK CANCER
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Months
Biospecimen Retention: Samples With DNA — blood, saliva, tissue.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patient with head and neck SCC: Anatomic location: oral cavity, larynx, oropharynx

SUMMARY:
Investigators have recently shown that epigenetic remodelling enzymes, such as HDAC inhibitors, are feasible drugs in HNC (8, 9). Preliminary data are indicating some deregulated epigenetics marks suggesting the corresponding histone modifiers as possible targets for the treatment of HNC, providing an attractive and feasible option to build upon. Our overarching hypothesis is that unique histone marks distinguish HPV+ and HPV- HNC and that specific histone modifiers are novel mediators of HNC tumorigenesis in an HPV specific manner

DETAILED DESCRIPTION:
Head and neck cancer (HNC) is a highly heterogeneous disease, involving diverse anatomical sites including oral cavity, larynx and oropharynx. HNC risk factors include tobacco smoking and alcohol consumption and, especially for the subtype of oropharyngeal cancers (OPC), human papillomavirus (HPV) infection

ELIGIBILITY:
Inclusion Criteria:• Age: Adults aged ≥ 18 years diagnosed with HNC

* Sex: Both male and female
* Human papilloma virus (HPV) test: Both positive and negative.
* Tumor: primary tumors, treatment naïve, squamous cell carcinoma
* Cancer stage: I-IV
* Anatomic location: oral cavity, larynx, oropharynx
* Tumor fragments not required for diagnostics

Exclusion Criteria:

* Previous radiotherapy, chemotherapy or immunotherapy for HNC
* Unable to provide written informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients that will undergo surgical tumor removal at the Otolaryngology - head and neck surgery unit of the IEO. Samples will be collected from at least 60 HNC primary tumors
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2024-03-06 (Actual); Primary Completion 2030-04-04 (Estimated); Study Completion 2030-04-04 (Estimated)

PRIMARY OUTCOMES:
PROFILING AND TARGETING EPIGENETIC MARKS TO IMPROVE DIAGNOSIS AND THERAPEUTIC APPROACHES IN HEAD AND NECK CANCER | 2 years
  define and fully characterize histone Post-Translational Modifications (hPTMs) and differentially expressed chromatin modifiers in HPV+ vs HPV- HNC through cutting-edge methodologies

CONTACTS AND LOCATIONS:
Overall Officials: Susanna Chiocca, Principal Investigator — Istituto Europeo di Oncologia
Locations (1):
- European Institute of oncology, Milan, MI, Italy